CLINICAL TRIAL: NCT02824237
Title: Bangladesh Center for Global Environmental and Occupational Health: A Study of Effects of Household Air Pollution on Cardio-pulmonary and Immune Function Outcomes Among Nonsmokers and Their Potential Prevention Avenues in Rural Bangladesh
Brief Title: GEOHealth Hub: Household Air Pollution and Cardio-pulmonary and Immune Function Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); National Institute of Environmental Health Sciences (NIEHS) (NIH); University of Chicago (Other); York University (Other); UChicago Research, Bangladesh (Unknown); Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other); Bangladesh Atomic Energy commission (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PR-15111; 1U01TW010120-01 (NIH)
Record Dates: First submitted 2016-06-28; First posted 2016-07-06 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Household Air Polution; Cardiovascular Diseases; Lung Diseases; Immune Dysfunction
MeSH Terms: conditions — Cardiovascular Diseases; Lung Diseases; Immune System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Improved cook stove (Experimental): The investigators will conduct a pre-post intervention study to evaluate effectiveness of improved stoves and compare outcomes after two years
  Interventions: Device: Improved cook stove

INTERVENTIONS:
Device: Improved cook stove — The investigators will conduct a pre-post intervention study to evaluate effectiveness of improved stoves and compare outcomes after two years

SUMMARY:
Background:

The increasing effect of environmental, occupational and climate change poses serious global threat for public health. More than half of the world's population, including around 85% people in Bangladesh, are exposed to household air pollutants (HAP). Environmental consequences of climate change are among the highest. Little evidence is available on the effects HAP on cardiopulmonary outcomes in low-income populations. Same is true for occupational health and climate change. The investigators will evaluate the effects of HAP on cardio-pulmonary and markers of immune function among non-smoking individuals. The investigators will also conduct two pilot studies to explore health effects associated with working in the garments industry and that of temperature due to climate changes.

Hypothesis:

1. Preclinical measures of cardiovascular diseases and pulmonary function are associated with exposure level of house hold air pollution (HAP) (assessed through PM2.5, CO and BC concentrations)
2. Stable biomarkers of immune function and inflammation are associated with exposure level of HAP.
3. Use of improved cook stove reduces exposure to HAP and thereby improve pre-clinical and molecular measures of cardio-pulmonary and immune functions.

Methods: The investigators will conduct a cross sectional study to assess the associations of HAP with preclinical makers of CVD among 600 non-smoking participants aged 25 to 65 years. Biomass exposure will be assessed for PM2.5, carbon Monoxide (CO) and black carbon (BC) by collecting personal air samples for 24-hour. Blood sample will be utilized from a subset of 200 adult participants and 60 children aged 3-5 years for assessing immune markers. The study will be conducted in icddr,b and URB study site at Matlab and Araihazar respectively.

After the cross sectional assessment, the investigators will conduct a pre-post intervention study to evaluate effectiveness of improved stoves in a subset of 200 homes. The investigators will measure the aforementioned markers after two years of cook stove installation. Finally, as pilot studies, health outcomes due to climate change (temperature change) and occupation (garment industry work) will be explored.

Outcome measures:

HAP will be assessed through PM2.5, CO and BC concentrations. Pulmonary function will be assessed through FEV1, FVC and FEV1/FVC. Preclinical makers of CVD will include RH-PAT, FMD, IMT, BAD, EKG and PFT. Markers of Immune function - proliferation of macrophage, dendritic cells (DC), neutrophils and T-cell, as well as macrophage derived cytokines (a panel of 17 or 27 cytokines) in peripheral blood mononuclear cells (PBMC)

ELIGIBILITY:
Inclusion Criteria:

1) aged between 25 and 65, 2) live in biomass using home with traditional stoves, 3) non-smoker and live with non-smokers, 4) exposed to <5 µg/L of water arsenic,

Exclusion Criteria:

1) Any immune related illness or taking any prescription medication (particularly those that suppress or enhance immune function), and 2) any clinical events of CVD or lung disease, including stroke or coronary heart disease.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
PM2.5 | Two Years
  The investigators will measure pre and post Changes in particulate matter <2.5 micrometers exposure (PM2.5) through 24-hour personal monitoring
CO | Two Years
  The investigators will measure pre and post Changes in carbon monoxide (CO) exposure through 24-hour personal monitors
FEV1 | Two Years
  The investigators will measure pre post changes in Forced Expiratory Volume in 1 second (FEV1) by spirometry
FVC | Two Years
  The investigators will measure pre post changes in Forced Vital Capacity (FVC) by spirometry
FEV1/FVC | Two Years
  The investigators will measure pre post changes in the ratio of Forced Expiratory Volume in 1 second and Forced Vital Capacity (FEV1/FVC) by spirometry
Reactive hyperemia-peripheral arterial tonometry (RH-PAT) (Endothelial dysfunction) | Two Years
  Endothelial dysfunction will be measured by reactive hyperemia-peripheral arterial tonometry (RH-PAT) and Pre and post comparison will be done pre post intervention changes will be assessed
Atherosclerosis [carotid intima-media thickness (cIMT)] | Two Years
  Atherosclerosis will be measured by ultrasound-assessed carotid intima-media thickness (cIMT) pre post intervention changes will be assessed
Vascular stiffness [brachial artery distensibility (BAD) ] | Two Years
  Vascular stiffness will be measured by brachial artery distensibility (BAD) and pre post intervention changes will be compared
Biomarkers of immune dysfunction and inflammation | Two Years
  Pre and post intervention changes of activation status of macrophages, dendritic cells and T-cell proliferation will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Yunus, MBBS, MSc., Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
All data collected of the proposed study will be made fully available to any bonafide researcher. In general, the investigators will follow the data sharing plan developed and practiced by the NIH-funded grantees. Any data request by external researchers will be reviewed by the PIs and the AOC and the requested specific data will be made available to the through a secured web-based interface developed specifically for this project. In general, data will be made available six months after the manuscript reporting results from those specific sets of data are accepted for publication and all data requests will be processed within six months from the receipt of the request in writing. Any data requests with potential conflicts will be reviewed and decided by the AOC.

REFERENCES:
- [Derived] Raqib R, Akhtar E, Ahsanul Haq M, Ahmed S, Haque F, Chowdhury MAH, Shahriar MH, Begum BA, Eunus M, Sarwar G, Parvez F, Sharker Y, Ahsan H, Yunus M. Reduction of household air pollution through clean fuel intervention and recovery of cellular immune balance. Environ Int. 2023 Sep;179:108137. doi: 10.1016/j.envint.2023.108137. Epub 2023 Aug 9. PMID 37579572